CLINICAL TRIAL: NCT01942213
Title: Observational Study to Evaluate and Compare the Rate and Extent of Inflammation After a Single Intravitreal Injection of Ranibizumab vs. a Single Intravitreal Injection of Aflibercept in Treatment Naive and Treatment Experienced Patients
Status: Completed | Type: Observational
Sponsor: Prism Vision Group (Other)
Responsible Party: Sponsor
Other Study IDs: NJRetina ML28942; NJRetina Observational ML28942 (Other: NJRetina); NCT01991730 (obsolete NCT alias)
Record Dates: First submitted 2013-09-10; First posted 2013-09-13 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Neovascular Age Related Macular Degeneration
Keywords: Macular; Degeneration; Age related; Neovascular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subjects receiving Ranibizumab: 150 Subjects diagnosed with Neovascular Age-Related Macular Degeneration receiving Ranibizumab 0.5 mg administered by intravitreal injection.
- Subjects receiving Aflibercept: 150 Subjects diagnosed with Age-related Macular Degeneration receiving Aflibercept 2 mg administered by intravitreal injection

SUMMARY:
This open-label, Phase IV prospective, observational study will evaluate patients, who have been diagnosed with Neovascular Age-Related Macular Degeneration and have previously received either a standard intravitreal injection of ranibizumab or aflibercept, in order to get and compare information regarding post-injection inflammatory (irritation in the eye)2-3 days post-injection.

Additionally, patients will be evaluated for visual acuity and pain 2-3 days post-injection.

DETAILED DESCRIPTION:
Patients, age 65 to 90, with Neovascular Age-Related Macular Degeneration who present for treatment with intravitreal ranibizumab or aflibercept will be selected in this study. 300 subjects from one site in the United States will be enrolled.

Inclusion Criteria:

* Ability to provide written informed consent and comply with study
* Age 65-90 years
* Diagnosis of Neovascular Age-Related Macular Degeneration who present for treatment with intravitreal ranibizumab or aflibercept

Exclusion Criteria:

* Previous intraocular inflammation
* Treatment with systemic anti-inflammatory agents
* Known systemic autoimmune diseases
* Treatment with intraocular steroids in the past 3 months
* History of intraocular surgery in the past 3 months
* Age greater than 90 years
* Patients who were switched between either therapies in the past 3 months

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age 65-90 years
* Diagnosis or Neovascular Age-Related Macular Degeneration who present for treatment with intravitreal ranibizumab or aflibercept

Exclusion Criteria:

* Previous intraocular inflammation
* Treatment with systemic anti-inflammatory agents
* Known systemic autoimmune diseases
* Treatment with intraocular steroids in the past 3 months
* History of intraocular surgery in the past 3 months
* Age greater than 90 years
* Patients who were switched between either therapies in the past 3 months

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Private practice patients referred to retinal specialist for treatment of Neovascular Age-Related Macular Degeneration
Sampling Method: Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2013-12; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
To evaluate post-intravitreal injection inflammatory response in patients receiving either ranibizumab or aflibercept. | 2-3 days after injection
  All eyes will be evaluated 2-3 days after injection and graded in terms of (a) aqueous cells, graded subjectively on a scale of 0-4, (b) aqueous flare, graded subjectively on a scale 0-4, (c) aqueous flare graded objectively with the FM-600 Kowa flare meter and (d) vitreous haze, graded subjectively on a scale of 0-4.

SECONDARY OUTCOMES:
To evaluate patients 2-3 days post-injection for best corrected visual acuity | 2-3 days post-injection
  Best corrected visual acuity will be assessed by the number of letters read correctly on the Early Treatment Diabetic Retinopathy Study eye chart at a starting test distance of 4 meters.

OTHER OUTCOMES:
To evaluate patient's pain post-injection | 2-3 days post-injection
  Pain will be measured on a standardized pain scale; Visual Function Questionaire -25 and a 0-10 numeric pain scale.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Roth, MD, Principal Investigator — Prism Vision Group
Locations (1):
- NJ Retina, Edison, New Jersey, United States